CLINICAL TRIAL: NCT04379271
Title: A Prospective, Multi-Center, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate the Efficacy, Safety and Tolerability of IMU-838 as Addition to Investigator's Choice of Standard of Care Therapy, in Patients With Coronavirus Disease 19
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of IMU-838 as Addition to Investigator's Choice of Standard of Care Therapy, in Patients With Coronavirus Disease 19 (COVID-19)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Immunic AG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2-IMU-838-COV
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, randomized, parallel-group trial
Who Masked: Participant, Investigator
Masking Description: Trial participants, the investigator and all other personnel directly involved in the conduct of the trial will be blinded to treatment assignments.
  To maintain the blind, IMU-838 and placebo tablets will have identical appearance, shape and color, and will have identical labeling and packaging. To minimize the potential for bias, treatment randomization information will be kept confidential by the responsible personnel and will not be released to investigators, other trial center personnel, or the Sponsor's designee(s).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMU-838 (Experimental): twice-daily (BID) oral 22.5 mg IMU-838 (45 mg/day + SoC)
  Interventions: Drug: IMU-838
- Placebo (Placebo Comparator): twice-daily (BID) oral placebo (+ SoC)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IMU-838 — Tablets will be taken BID with a glass of water (if possible); one tablet each in the morning (15 to 50 min before a meal if applicable), and in the evening (2 hours after any meal if applicable).
  If the patient is intubated for ventilation, IMP is to be given via a gastric tube. The tablet has no coating and a homogeneous content and can be crushed into smaller pieces (if necessary) for dosing via gastric tube.
  Other Names: vidofludimus calcium
  Arms: IMU-838
Other: Placebo — Matching placebo, twice-daily administration BID as described for the test product, identical number of tablets as given for IMU-838
  Arms: Placebo

SUMMARY:
At present there is no approved drug treatment for Covid-19. In this study we plan to investigate if an experimental drug called IMU-838 (vidofludimus calcium) can improve your symptoms, prevent worsening that would initiate further treatments such as ventilation, and can lower your virus number if given in addition to your doctor's choice of standard therapy. We will also test if IMU-838 has any side effects and measure the level of IMU 838 in your blood.

Experimental drug means that it is not yet authorized for marketing in your country. To date approximately 600 individuals have received IMU-838 (or a drug similar to IMU-838 that contains the same active substance as IMU-838) in research studies.

DETAILED DESCRIPTION:
The trial consists of a Phase 2 proof-of-concept phase (Part 1) with the option to extend enrollment (without interruption) to Phase 3 (Expansion Phase, Part 2).

This trial is a multicenter, double-blind, placebo-controlled, randomized, parallel-group trial to evaluate the safety and efficacy of IMU-838 as addition to investigator's choice of SoC treatment in patients with COVID-19. Eligible patients will be centrally randomized 1:1 to twice-daily (BID) oral 22.5 mg IMU-838 (45 mg/day + SoC) or placebo (+ SoC). Randomization will be stratified by age (< or >=65 years) and antiviral therapy (no antivirals, Hydroxychloroquine and Chloroquine, all other antivirals).

Adaptive sequential trial design and overall trial design

The trial uses an adaptive sequential design. An IDMC will review unblinded data and provide the Sponsor with recommendations regarding modifications of sample size and trial conduct.

A 1st interim analysis (IA1) will be performed after approximately 200 patients have completed the trial (either as scheduled or prematurely), while enrollment continues. If no activity of IMU 838 is observed by the IDMC in this IA, further patient enrollment will be stopped, and a final analysis of Part 1 will be performed (FA1). It is expected that the final analysis of Part 1 will include approximately 230 patients. If the IA1 results indicate activity of IMU-838 in COVID-19, the trial may be extended to Part 2 with a revised sample size derived by the IDMC based on IA1 results and with possible other trial adjustments. If the trial is extended into Part 2, a 2nd IA (IA2) is planned after approximately two-thirds of patients (based on the overall global sample size [Part 1 and Part 2 combined]) have been enrolled to potentially adjust sample size and other trial features if needed. The final analysis of the trial (FA2) will then be done after all patients have completed Part 2.

In addition, an early interim safety analysis will be performed and evaluated by the IDMC after 30 patients have been enrolled to assess unblinded safety data. Further safety analyses can be initiated at any time by the IDMC or Sponsor when new safety signals are identified within this or other trials of IMU-838.

Screening

Patients can be screened for a maximum of 2 days (from Day -2 to Day 0) and eligible patients will be randomized on Day 0 and treated with IMP + SoC for 14 days. It is encouraged to screen potential participants immediately at the day of hospitalization (including informed consent, assessment of inclusion/exclusion criteria, screening laboratory tests all done locally, assessment of clinical and blood gas criteria) and randomize patients on the same day (Day 0). To assess eligibility criteria, existing local laboratory values obtained within 48 hours of randomization can also be used, except for testing of positive status of SARS-CoV-2 infection where a 4-day window is allowed.

IMP administration should start as quickly as possible after randomization and first IMP intended to be given in the evening of the screening day (Day 0).

Blinded Treatment period (Day 0 to Day 13) and Day 14 (end-of-treatment)

The first dose of IMP (2 tablets) should always be given on Day 0 (allowed range for first dose: 12:00 noon on Day 0 to 02:00 a.m.). All further IMP doses are 1 tablet each in the morning and evening. Information about the status and patient care are continuously obtained and documented once or twice daily.

After the last IMP dose in the evening of Day 13, the end-of-treatment assessments will be done on Day 14. Blood sampling for IMU-838 trough values must be performed in the morning around the time the morning dose was usually taken by the respective patient. Patients may then continue to receive SoC without any further restrictions on concomitant medications as during the 14-day BT period .

Day 28 Visit (EoS)

The patient should return for the final trial visit on Day 28 (EoS). If IMP is prematurely discontinued for any reason, the EoS visit should always be conducted on Day 28 and no earlier EoS should be performed. If patients withdraw from IMP prematurely, they should be encouraged to allow the EoS visit as part of the follow-up. If the patient dies during the trial, the investigator should indicate that this visit was not performed. However, even if no EoS visit was performed, information about patient status should be reported on the EoS page in the case report form. If the patient refuses any EoS visit or the patient is lost to follow-up, it is permissive in this trial that the investigator contacts the patient, the family of the patient or the referring physician by phone or email to obtain status of life information, or is able to search in registers or publicly available information for such status of life information.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years old (may be extended to include also children 12 years or older after the 1st interim analysis)
2. Admitted to the hospital or other medical in-patient treatment facility for treatment of COVID-19 The hospitalization needs to be for medical reasons (treatment of COVID-19 disease) and cannot be for social reasons or due to housing insecurity.

   For US sites only: If the investigator would commonly hospitalize the patient but for healthcare resource reasons decides to treat the patient in a specially designed out-patient setting, then such patients are also allowed to enter the trial (please note that in this case the patient would be counted as clinical status category 3). The investigator then must assure that the patient has at least a twice daily assessment by qualified trial personnel and all laboratory assessments can be adequately performed as per protocol. The Sponsor reserves the right to discontinue this option via administrative letter if such assurances cannot be met by any site.
3. SARS-CoV-2 infection confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) test in a nasopharyngeal, oropharyngeal or respiratory sample at ≤4 days before randomization
4. Moderate COVID-19 disease defined as fulfilling clinical status category 3 or 4 on the WHO 9-point ordinal scale [21]:

   * Category 3: Hospitalized (see note above for US only), virus-positive, no oxygen therapy with the following conditions:
   * The hospitalization needs to be for medical reasons (treatment of COVID-19 disease) and cannot be for social reasons or due to housing insecurity
   * Category 4: Hospitalized, virus-positive, oxygen by mask or nasal prongs (excluding high-flow oxygen therapy) with the following conditions:
   * Peripheral capillary oxyhemoglobin saturation (SpO2) >92% at maximum of 6 liters oxygen flow per minute
   * Stable respiratory rate ≤30 breaths/min at maximum of 6 liters oxygen flow per minute
5. Presence of at least 1 symptom characteristic for COVID-19 disease i.e., fever, cough or respiratory distress
6. Willingness and ability to comply with the protocol
7. Written informed consent given prior to any trial-related procedure
8. For women of childbearing potential: Application of a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly) together with a barrier method between trial consent and 30 days after the last intake of the IMP.

   Highly effective forms of birth control are those with a failure rate less than 1% per year and include:
   * oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraceptives associated with inhibition of ovulation
   * oral, injectable, or implantable progestogen-only hormonal contraceptives associated with inhibition of ovulation
   * intrauterine device or intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * vasectomized partner (i.e., the patient's male partner underwent effective surgical sterilization before the female patient entered the clinical trial and is the sole sexual partner of the female patient during the clinical trial)
   * sexual abstinence (acceptable only if it is the patient's usual form of birth control/lifestyle choice; periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are no acceptable methods of contraception)

   Barrier methods of contraception include:
   * Condom
   * Occlusive cap (diaphragm or cervical/vault caps) with spermicidal gel/film/cream/suppository
9. Male patients must agree not to father a child or to donate sperm starting at Screening, throughout the clinical trial and for 30 days after the last intake of the IMP. Male patients must also

   * abstain from sexual intercourse with a female partner (acceptable only if it is the patient's usual form of birth control/lifestyle choice), or
   * use adequate barrier contraception during treatment with the IMP and until at least 30 days after the last intake of the IMP, and
   * if they have a female partner of childbearing potential, the partner should use a highly effective contraceptive method as outlined in inclusion criterion 8
   * if they have a pregnant partner, they must use condoms while taking the IMP to avoid exposure of the fetus to the IMP

Exclusion Criteria:

Underlying disease-related exclusion criteria

1. Involvement in the trial is not in the patient's best interest according to the investigator's decision, including the presence of any condition that would, in the assessment of the investigator, not allow the protocol to be followed safely Note: The investigator should particularly consider exclusion of patients at increased risk for serious or fatal AEs in case of worsening of the pulmonary perfusion. This includes, but is not limited to, pre-existing pulmonary hypertension, severe chronic respiratory disease, severely increased risk for thromboembolic complications and moderate to severe left ventricular ejection fraction (LVEF) dysfunction. In addition, other known risk factors of highest risk of mortality in COVID-19 patients should be considered.
2. Presence of respiratory failure, shock, and/or combined failure of other organs that requires ICU monitoring in the near foreseeable future
3. Critical patients whose expected survival time <48-72 hours
4. Presence of the following laboratory values at screening:

   * White blood cell count (WBC) <1.0 x 109/L
   * Platelet count <100,000/mm³ (<100 x 109/L)
   * Total bilirubin>2 x ULN
   * Alanine aminotransferase (ALT) or gamma glutamyl transferase (GGT) >5 x ULN
5. Participation in any other interventional clinical trial
6. Hospitalization primarily for other reasons than COVID-19 (including primarily for concomitant conditions during ongoing SARS-CoV-2 infection)
7. Anticipated transport to a different hospital or institution, in particular when such transport is anticipated for pending ECMO or RRT treatment
8. Clinical suspicion of a bacterial superinfection at Screening IMP-related exclusion criteria
9. Patients who cannot take drugs orally
10. Allergic or hypersensitive to the IMP or any of the ingredients
11. Use of the following concomitant medications is prohibited from Screening to end of treatment with IMP in this trial (up to Day 14) if not indicated otherwise in this protocol:

    * Concurrent use of any mycophenolate mofetil or of methotrexate exceeding 17.5 mg weekly
    * Any medication known to significantly increase urinary elimination of uric acid, in particular lesinurad (Zurampic™) as well as uricosuric drugs such as probenecid
    * Current treatments for any malignancy, in particular irinotecan, paclitaxel, tretinoin, bosutinib, sorafenib, enasidenib, erlotinib, regorafenib, pazopanib and nilotinib
    * Any drug significantly restricting water diuresis, in particular vasopressin and vasopressin analogs
    * Use of rosuvastatin at daily doses higher than 10 mg
    * Arbidol and Colchicine
    * Any use of other DHODH inhibitors, including teriflunomide (Aubagio™) or leflunomide (Arava™)
    * Chloroquine and Hydroxychloroquine during the entire trial unless taken for indicated use before entering the trial
12. Use of any investigational product within 8 weeks or 5x the respective half-life before the date of informed consent, whichever is longer, and throughout the duration of the trial General exclusion criteria
13. Patients who have a "do not intubate" or "do not resuscitate" order (unless the patient waives in writing this order and will allow intubation for the duration of the trial period)
14. Patients with end-stage liver disease (Child Pugh C score)
15. History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (New York Heart Association [NYHA] class 3 or 4) Note: NYHA class 3: Cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. NYHA class 4: Cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
16. Legal incapacity, limited legal capacity, or any other condition that makes the patient unable to provide consent for the trial
17. Pregnant or breastfeeding
18. An employee of an investigator or Sponsor or an immediate relative of an investigator or Sponsor
19. Patients institutionalized due to judicial order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Bulgaria (2):
  - Military Medical Academy, Clinic of Infectious Diseases, Sofia
  - UMHATEM N.I.Pirogov, Clinic of internal diseases, Sofia
- Germany (2):
  - University Hospital Frankfurt, Infectious Diseases, Frankfurt
  - Clinic of the Hannover Medical School, Pneumology Clinic, Hanover

REFERENCES:
- [Derived] Vehreschild MJGT, Atanasov P, Yurko K, Oancea C, Popov G, Smesnoi V, Placinta G, Kohlhof H, Vitt D, Peelen E, Mihajlovic J, Muehler AR. Safety and Efficacy of Vidofludimus Calcium in Patients Hospitalized with COVID-19: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Trial. Infect Dis Ther. 2022 Dec;11(6):2159-2176. doi: 10.1007/s40121-022-00690-0. Epub 2022 Oct 15. PMID 36242741

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 223 patients were randomized; 220 patients were treated and included in the full analysis and safety data set (110 patients each in the 45 mg IMU-838 group and the placebo group).
Groups:
- IMU-838: twice-daily (BID) oral 22.5 mg IMU-838 (45 mg/day + SoC)
  IMU-838: Tablets will be taken BID with a glass of water (if possible); one tablet each in the morning (15 to 50 min before a meal if applicable), and in the evening (2 hours after any meal if applicable).
  If the patient is intubated for ventilation, IMP is to be given via a gastric tube. The tablet has no coating and a homogeneous content and can be crushed into smaller pieces (if necessary) for dosing via gastric tube.
Period: Overall Study
Arm/Group | IMU-838 | Placebo
Started | 110 | 110
Completed | 93 | 97
Not Completed | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMU-838 | Placebo | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 83 | 166
  >=65 years | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.4) | 53.7 (14.2) | 54.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 46 | 101
  Male | 55 | 64 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 110 | 107 | 217
  Race: Asian | 0 | 1 | 1
  Race: Black or African American | 0 | 1 | 1
  Race: Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without Any Need for INV Until EoS
Description: Number of Participants Stratified as those With and Without the Need for INV Until End-of-study (EoS). For this outcome a worst case approach was used in which patients who were lost to follow-up or who discontinued the trial on or before Day 13 due to any other reason than death and discontinued with a last observed WHO clinical status no lower than that at Screening, and patients who died were considered as patients requiring INV.
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: FAS, Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants
  No INV needed | 98 | 101
  INV needed | 12 | 9

2. Secondary Outcome: Days in ICU Department
Description: Duration of ICU Treatment Until EoS for Only Patients Who Were Admitted to the ICU During the Trial.
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 4 | 5
days | 2.54 (7.24) | 2.33 (7.24)

3. Secondary Outcome: All Cause Mortality (ITT Approach)
Description: 28-day All-cause Mortality (including lost to follow-up): 'all-cause-mortality' includes all confirmed deaths and patients who discontinued the trial before Day 28 and for whom no outcome (alive or dead) could be determined at EoS; 'actual death' includes only those patients for which a fatal outcome was confirmed by Day 28.
Time Frame: Throughout the Study (Day 0 to Day 28 )
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants
  actual death | 2 | 2
  28 days all cause mortality (including lost to follow-up) | 9 | 8

4. Secondary Outcome: Time to Clinical Improvement
Description: Defined as the time from first dose of investigational medicinal product (IMP) to an improvement of at least 2 points on the Modified WHO Ordinal Scale for Clinical Status (Modified WHO Ordinal Scale for Clinical Status), or live discharge from hospital without oxygen supplementation, whichever comes first. The 50% Kaplan-Meier quartile (median) of actual values per treatment arm is provided as outcome of this variable below.
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
days | 13.70 [13.70 to 13.80] | 13.80 [13.70 to 13.80]

5. Secondary Outcome: Days of Hospitalization
Description: Duration of hospitalization (for US sites only: or treatment in special outpatient setting in lieu of hospitalization due to resource restraints)cacy:
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: Patients from Bulgaria were excluded because they had to stay in hospital for the entire treatment period as per protocol.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 73 | 77
days | 13.49 (7.00) | 14.35 (7.71)

6. Secondary Outcome: Patients Free of Renal-replacement Therapy (RRT)* Until EoS
Description: Number of Patients Both for All Patients and Surviving Patients Free of Renal-replacement Therapy (RRT)* Until EoS
Time Frame: Throughout the Study (Day 0 to Day 28 )
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants | 110 | 110

7. Secondary Outcome: Patients Required ECMO Until EoS
Description: Number and Percentage of patients both for all patients and surviving patients free from extracorporeal membrane oxygenation (ECMO)* until EoS.
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: If ECMO was prescribed but was not started, the patient is considered as being not free of ECMO.
  Patients with ECMO documented are included with 'no' in analysis of all following visits (irrespective of whether visit was done). Patients without ECMO documented are excluded from analysis of visits after their last performed visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants | 0 | 0

8. Secondary Outcome: Patients Free of INV Until Day 14*
Description: Number and persentage of patients free of INV until Day 14*
Time Frame: Throughout the Study (Day 0 to Day 14 )
Population: Patients without INV documented in group IMU-838 and Placebo group ( 7 and 10 accordingly) were excluded from analysis of visits after their last performed visit
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 103 | 100
Participants | 102 | 99

9. Secondary Outcome: Patients Free of RRT
Description: Percentage of patients free of RRT until Day 14*
Time Frame: Day 0 to Day 14
Population: Patients without RRT documented are excluded from analysis of visits after their last performed visit.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants | 110 | 110

10. Secondary Outcome: Number of Patients Free of ECMO
Description: Number of patients free of ECMO until Day 14.
Time Frame: Day 0 to Day 14
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants | 110 | 110

11. Secondary Outcome: Patients With Improvement of at Least 2 Points (From Randomization) on the 9-category WHO Ordinal scale1
Description: Numbers of patients with improvement of at least 2 points (from randomization) on the 9-category WHO ordinal scale1( Modified WHO Ordinal Scale for Clinical Status)on Days 6, 14, and 28, where score 0 means no clinical or virological evidence of infection and score 8 is the worth outcome ( mens death).
Time Frame: on Days 6, 14, and 28
Measure: Number; unit: participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
participants
  Day 6 | 5 | 5
  Day 14 | 44 | 39
  Day 28 | 95 | 93

12. Secondary Outcome: Patients With Auxiliary Oxygen Therapy (Including All Types of Oxygen Therapy)
Description: Percentage of Patients with auxiliary oxygen therapy (including all types of oxygen therapy) on Days 6, 14, and 28.
Time Frame: on Days 6, 14, and 28
Population: Patients without axillary oxygen therapy documented were excluded from analysis of visits after their last performed visit. Numbers of participants analyzed changed across time points.
Measure: Number; unit: percentage of participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 108 | 108
percentage of participants
  Day 6 | 47.2 | 40.7
  Day 14: number analyzed (Participants) | 107 | 107
  Day 14 | 47.7 | 41.1
  Day 28: number analyzed (Participants) | 106 | 107
  Day 28 | 48.1 | 42.1

13. Secondary Outcome: Patients With Clinical Recovery
Description: Percentage of Patients With Clinical Recovery: Axillary Temp <= 36.6 °C, or Oral Temp <= 37.2 °C, or Rectal or Tympanic Temp <= 37.8 °C and Respiratory Frequency <= 24 Times/Min Without O2 Inhalation and O2 Saturation >= 98% Without O2 Inhalation
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: Clinical recovery was only assumed if it was confirmed in the evening and at the next visit.
Measure: Number; unit: percent of patients
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 109 | 110
percent of patients
  Baseline | 3.7 | 3.6
  Day 0 | 5.5 | 3.7
  Day 7 | 17.4 | 12.0
  Day 10 | 21.7 | 19.5
  Day 14 | 40.2 | 45.8
  Day 28 | 69.3 | 65.6

14. Secondary Outcome: Patients With Clinical Recovery
Description: Percentage of Patients With Clinical Recovery Oxygen Saturation ≥98% Without Oxygen Inhalation
Time Frame: Throughout the Study (Day 0 to Day 28 )
Measure: Number; unit: percent of patients
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 103 | 103
percent of patients
  Day 7 | 17.4 | 12.0
  Day 14 | 40.2 | 45.8
  Day 28 | 69.3 | 65.6

15. Secondary Outcome: Patients With Clinical Improvement or Live Discharge From Hospital Without Oxygen Supplementation
Description: Percentage of patients with clinical improvement, defined as the time from first dose of IMP to an improvement of at least 2 points on the WHO 9 category ordinal scale, or live discharge from hospital without oxygen supplementation, whichever comes first (Modified WHO Ordinal Scale for Clinical Status, where score 0 - for patient with no clinical or virological evidence of infections, score 9 - the worth scenario- death)
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: One patient from group IMU-838 was excluded from this analysis due to hospital discharge before start of treatment.
Measure: Number; unit: percent of patients
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 109 | 110
percent of patients | 91.7 | 88.2

16. Secondary Outcome: Percentage of Participants With WHO Status<=2
Description: Clinical patient status on the 9-category WHO ordinal scale1 on Days 6, 14, and 28
Time Frame: on Days 6, 14, and 28
Population: Missing data
Measure: Number; unit: percentage of patients, WHO status <=2
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
percentage of patients, WHO status <=2
  Day 6: number analyzed (Participants) | 95 | 98
  Day 6 | 6.3 | 5.1
  Day 14: number analyzed (Participants) | 99 | 83
  Day 14 | 48.5 | 44.3
  Day 28: number analyzed (Participants) | 97 | 100
  Day 28 | 97.9 | 96.9

17. Secondary Outcome: Duration of INV
Description: Duration of INV throughout the study. If no entry on the respective CRF page exists, the duration is set to 0 days for patients who performed Day 28 visit. Patients without Day 28 visit and without any entry on the respective CRF page are excluded from analysis.
Time Frame: Throughout the Study (Day 0 to Day 28 )
Population: Patients who are lost to follow-up or discontinued the trial on or before Day 13 (last treatment day) due to any other reason than death and discontinue with a last observed WHO clinical status, and patients who die before Day 28 will be considered treatment failures (i.e. having a need for INV) for the primary endpoint.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 99 | 100
days | 0.00 [0 to 0.1] | 0.07 [0 to 7.0]

18. Secondary Outcome: Days on ECMO
Description: Duration of ECMO in days (duration set to 0 for those who did not require ECMO). No participants required ECMO.
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: patients, who require ECMO throughout the study
Measure: Number; unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
days | 0 | 0

19. Secondary Outcome: Days on RRT
Description: Duration of RRT in days (duration set to 0 for those who did not require RRT).No participants required RRT.
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: patients , who require RRT throughout the study
Measure: Number; unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
days | 0 | 0

20. Secondary Outcome: Days of Auxiliary Oxygen Therapy
Description: Duration of auxiliary oxygen therapy (including all types of oxygen therapy)
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: 106 and 107 participants respectively were studied. Only participants who required auxiliary oxygen therapy were selected. If auxiliary oxygen therapy started before randomization, time of randomization is used as start time.Patients who are lost to follow-up or discontinue prematurely without Day 28 and without any auxiliary oxygen therapy documented are excluded from analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 51 | 45
days | 4.49 (7.01) | 3.86 (7.26)

21. Secondary Outcome: Days of Hospitalization
Description: Duration of hospitalization for survivors
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: Patients enrolled in centers in Bulgaria (N = 37 in the 45 mg IMU-838 group and N = 33 in the placebo group) were excluded from the analysis as, per protocol, they were required to remain hospitalized for the entire treatment period
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 71 | 75
days | 13.53 [6.90 to 15.90] | 14.52 [7.30 to 19.00]

22. Secondary Outcome: Participants With ICU Admission
Description: Percentage of Participants with ICU Admission at different time point
Time Frame: on Days 6, 14, and 28
Population: Patients without ICU documented were excluded from analysis of visits after their last performed visit.
Measure: Number; unit: percent of patients
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 107 | 105
percent of patients
  Day 6 | 3.7 | 3.8
  Day 14 | 3.8 | 5.0
  Day 28 | 4.0 | 5.0

23. Secondary Outcome: Probability of Death
Description: Probability of death derived from Kaplan Meier analyses
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Number; unit: Probability
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Probability | 0.019 | 0.019

24. Secondary Outcome: Days to INV
Description: Time to first prescription of invasive ventilation (INV). The time to first prescription of INV, only patients with actual INV or prescription for INV are considered.
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: Only 2 patients had confirmed use of INV throughout the study and were included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 1 | 1
days | 13.8 [13.8 to 13.8] | 6.0 [6.0 to 6.0]

25. Secondary Outcome: Days to RRT
Description: Time to first prescription of RRT
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: No patients required RRT during the trial
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Days to ECMO
Description: Time to first prescription of ECMO
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: No patients required ECMO during the trial
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Days to INV, RRT and ECMO
Description: Time to first prescription of INV, RRT, and ECMO. The time to first prescription of INV, only patients with actual INV or prescription for INV are considered.
Time Frame: Throughout the Study (Day 0 to Day 28)
Population: Only 2 patients had confirmed use of INV throughout the study and were included in the analysis. No patients required RRT or ECMO during the trial.
Measure: Median (Full Range); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 1 | 1
days | 13.8 [13.8 to 13.8] | 6.0 [6.0 to 6.0]

28. Secondary Outcome: Probability of ICU Admission
Description: Overall probability of ICU admission derived from Kaplan Meier analyses.
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Number; unit: Probability
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Probability | 0.037 | 0.047

29. Secondary Outcome: Cumulative Dose
Description: Cumulative Dose of Vasoactive Therapies and Days With Vasoactive Therapies (Daily Until Day 14)
Time Frame: Day 0 to day 14
Population: Vasoactive therapy was prescribed for only 1 patient in the IMU-838 group for a single day . If no vasoactive therapy was given, cumulative dose is set to 0.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IMU-838
Number analyzed (Participants) | 1
mg | 0

30. Secondary Outcome: Time to Clinical Recovery
Description: Time of first assessments of parameters contributing to clinical recovery
Time Frame: Throughout the Study (Day 0 to EoS [Day 27 up to Day 42])
Population: The first clinical recovery is counted when later relapses are absent. Except for Day 28/early termination/last day with non-missing assessment, only events where clinical recovery is confirmed on the next visit with non-missing assessment(s) are counted. For Day 28/early termination/last day with non-missing assessment this confirmation is not needed. EoS can be > 28 days as due to COVID-19 restrictions some patients came late (up to Day 42), which was considered a minor protocol deviation.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
days | 14.10 [12.90 to 27.80] | 14.10 [13.70 to 27.90]

31. Secondary Outcome: Plasma Levels of IMU-838
Description: Morning trough plasma levels of IMU-838 on Days 0, 1, 2, 3, 6, 14, and 28
Time Frame: on Days 0, 1, 2, 3, 6, 14, and 28
Population: Placebo group not available
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | IMU-838
Number analyzed (Participants) | 110
ug/mL
  Baseline | 0.1108 (0.1135)
  Day 1 | 2.9234 (1.1493)
  Day 2 | 3.5724 (1.6299)
  Day 3 | 3.8572 (1.8606)
  Day 6 | 4.3607 (2.4872)
  Day 14 | 4.6514 (2.6506)
  Day 28 | 0.1014 (0.0093)

32. Secondary Outcome: Correlation of Trough Levels (Quartiles) to Selected Clinical Outcomes
Description: Kaplan-Meier analyses were used to investigate a potential relationship between trough plasma levels of IMU-838 and time to clinical improvement and time to clinical recovery. Estimates of the clinical outcomes were evaluated separately for patients within each of the four quartiles of IMU-838 trough levels at Day 14.
Time Frame: Trough levels at Day 14; Clinical outcome: Day 0 to EoS (EoS = Day 27 up to Day 42)
Population: The safety analysis set consisting of all randomized patients who received at least one dose of IMU-838.
Measure: Median (90% Confidence Interval); unit: days
Groups:
- IMU-838: 110 participants analyzed, who received twice-daily (BID) oral 22.5 mg IMU-838 (45 mg/day + SoC)
  IMU-838: Tablets will be taken BID with a glass of water (if possible); one tablet each in the morning (15 to 50 min before a meal if applicable), and in the evening (2 hours after any meal if applicable).
  If the patient is intubated for ventilation, IMP is to be given via a gastric tube. The tablet has no coating and a homogeneous content and can be crushed into smaller pieces (if necessary) for dosing via gastric tube.
Arm/Group | IMU-838
Number analyzed (Participants) | 94
days
  Time to clinical recovery - Q1 (Min to 3.1 µg/mL IMU-838): number analyzed (Participants) | 24
  Time to clinical recovery - Q1 (Min to 3.1 µg/mL IMU-838) | 27.8 [13.2 to 29.1]
  Time to clinical recovery - Q2 (3.1 to 4.2 µg/mL IMU-838): number analyzed (Participants) | 23
  Time to clinical recovery - Q2 (3.1 to 4.2 µg/mL IMU-838) | 27.9 [12.9 to 28.8]
  Time to clinical recovery - Q3 (4.2 to 6.0 µg/mL IMU-838): number analyzed (Participants) | 24
  Time to clinical recovery - Q3 (4.2 to 6.0 µg/mL IMU-838) | 11.8 [6.0 to 13.7]
  Time to clinical recovery - Q4 (6.0 µg/mL to Max IMU-838): number analyzed (Participants) | 23
  Time to clinical recovery - Q4 (6.0 µg/mL to Max IMU-838) | 11.3 [4.8 to 14.1]
  Time to clinical improvement - Q1 (Min to 3.1 µg/mL IMU-838): number analyzed (Participants) | 24
  Time to clinical improvement - Q1 (Min to 3.1 µg/mL IMU-838) | 13.7 [13.7 to 14.0]
  Time to clinical improvement - Q2 (3.1 to 4.2 µg/mL IMU-838): number analyzed (Participants) | 23
  Time to clinical improvement - Q2 (3.1 to 4.2 µg/mL IMU-838) | 13.8 [13.7 to 14.8]
  Time to clinical improvement - Q3 (4.2 to 6.0 µg/mL IMU-838): number analyzed (Participants) | 24
  Time to clinical improvement - Q3 (4.2 to 6.0 µg/mL IMU-838) | 13.7 [13.1 to 13.8]
  Time to clinical improvement - Q4 (6.0 µg/mL to Max IMU-838): number analyzed (Participants) | 23
  Time to clinical improvement - Q4 (6.0 µg/mL to Max IMU-838) | 13.7 [11.0 to 13.9]

33. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: Adverse events (AEs) and serious AEs. AEs-Hypertriglyceridemia,Increased glycosylated hemoglobin, Headache, Thrombocytosis, Hyperglycemia, AEs reported in ≥ 2.0% of patients in any treatment group included anemia, bradycardia, sinus bradycardia, tachycardia, pyrexia, hepatocellular injury, hematuria, hypertension and hypertensive crisis. SAEs- deep vein thrombosis,COVID-19 pneumonia, patient death.
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants
  Any AE | 81 | 69
  Any serious AE | 2 | 4

34. Secondary Outcome: Vital Signs: Height
Description: Safety Height in centimeters will be recorded without shoes. Changes in vital signs judged by the investigator as clinically significant will be reported as an AE.
Time Frame: at Baseline
Population: For 55 female and 55 male in group IMU-838 and 46 female and 64 male in Placebo group
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- IMU-838: For 55 female and 55 male in this group: twice-daily (BID) oral 22.5 mg IMU-838 (45 mg/day + SoC)
  IMU-838: Tablets will be taken BID with a glass of water (if possible); one tablet each in the morning (15 to 50 min before a meal if applicable), and in the evening (2 hours after any meal if applicable).
  If the patient is intubated for ventilation, IMP is to be given via a gastric tube. The tablet has no coating and a homogeneous content and can be crushed into smaller pieces (if necessary) for dosing via gastric tube.
- Placebo: For 46 female and 64 male in this group: twice-daily (BID) oral placebo (+ SoC)
  Placebo: Matching placebo, twice-daily administration BID as described for the test product, identical number of tablets as given for IMU-838
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
centimeters
  Male: number analyzed (Participants) | 55 | 64
  Male | 178.1 (5.7) | 175.6 (6.8)
  Female: number analyzed (Participants) | 55 | 46
  Female | 163.0 (5.5) | 163.9 (4.4)

35. Secondary Outcome: Vital Signs: Weight
Description: Safety Weight in kilograms will be recorded without shoes. Changes in vital signs judged by the investigator as clinically significant will be reported as an AE.
Time Frame: at Baseline
Population: For 55 female and 55 male in group IMU-838 and 46 female and 64 male in Placebo group.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
kilograms
  Male: number analyzed (Participants) | 55 | 64
  Male | 92.98 (18.86) | 88.95 (14.05)
  Female: number analyzed (Participants) | 55 | 46
  Female | 77.88 (14.46) | 74.09 (13.89)

36. Secondary Outcome: Vital Signs: Body Temperature (ºC)
Description: Safety Body temperature can be measured axillary, oral, rectal or tympanic, but should be always measured by the same method for a patient. Changes in vital signs judged by the investigator as clinically significant will be reported as an AE.
Time Frame: at Baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 108 | 109
degrees Celsius | 36.86 (0.58) | 36.75 (0.53)

37. Secondary Outcome: Albumin Concentration at Various Time Points
Description: Clinical laboratory parameters: blood chemistry (Albumin concentration at various time points)
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 108
g/L
  Baseline | 39.4 (4.4) | 40.2 (4.7)
  Day 6 | 37.9 (4.2) | 38.7 (4.9)
  Day 14 | 39.6 (4.6) | 40.3 (4.6)
  Day 28 | 44.0 (3.7) | 44.0 (4.4)

38. Secondary Outcome: Hematocrit Ratio at Various Time Points
Description: Clinical laboratory parameters: hematology- Hematocrit ratio at various time points
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 108 | 106
ratio
  Baseline | 0.435 (0.052) | 0.448 (0.053)
  Day 6 | 0.430 (0.059) | 0.443 (0.053)
  Day 14 | 0.435 (0.049) | 0.440 (0.051)
  Day 28 | 0.428 (0.046) | 0.432 (0.052)

39. Secondary Outcome: Urine Creatinine at Various Time Points
Description: Clinical laboratory parameters: urinalysis- Urine creatinine at various time points
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 109 | 107
umol/L
  Baseline | 11368.1 (7672.0) | 11303.9 (6496.6)
  Day 6 | 9259.5 (5198.1) | 10214.0 (6551.3)
  Day 14 | 8940.8 (5771.0) | 10040.1 (6399.2)
  Day 28 | 10498.2 (7776.1) | 11589.2 (6665.9)

40. Secondary Outcome: Temperature
Description: Temperature data at different time point.
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 108 | 109
degrees Celsius
  Baseline | 36.9 (0.58) | 36.8 (0.53)
  Day 6 | 36.7 (0.33) | 36.5 (0.42)
  Day 14 | 36.4 (0.24) | 36.4 (0.34)
  Day 28 | 36.4 (0.21) | 36.4 (0.34)

41. Secondary Outcome: D-dimer
Description: Disease markers
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 109
ng/mL
  Baseline | 529.5 [79 to 19520] | 473.0 [106 to 5647]
  Day 14 | 348.0 [91 to 19520] | 357.0 [60 to 19520]
  Day 28 | 343.0 [100 to 19520] | 332.5 [76 to 9076]

42. Secondary Outcome: Lactate Dehydrogenase (LDH)
Description: Blood levels of disease markers
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (Full Range); unit: nkat/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
nkat/L
  Baseline | 4176.0 [1900 to 14886] | 4059.0 [1900 to 14886]
  Day 14 | 3167.0 [1650 to 11302] | 3117.0 [1850 to 10752]
  Day 28 | 3375.5 [1650 to 7918] | 3267.0 [1650 to 15053]

43. Secondary Outcome: C-reactive Protein
Description: Blood levels of disease markers
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (Full Range); unit: nmol/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
nmol/L
  Baseline | 320.4826 [5.7144 to 2682.911] | 245.2430 [5.7144 to 2362.904]
  Day 14 | 27.61960 [5.7144 to 6328.698] | 20.95280 [5.7144 to 858.1124]
  Day 28 | 23.81000 [5.7144 to 207.6232] | 16.19080 [5.7144 to 1447.648]

44. Secondary Outcome: Troponin I
Description: Bood levels of disease markers
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (Full Range); unit: ug/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 103 | 97
ug/L
  Baseline | 0.00860 [0.0086 to 0.0904] | 0.00860 [0.0086 to 0.1054]
  Day 14 | 0.00860 [0.0086 to 0.0812] | 0.00860 [0.0086 to 1.0152]
  Day 28 | 0.00860 [0.0086 to 0.0542] | 0.00860 [0.0086 to 0.1053]

45. Secondary Outcome: Procalcitonin
Description: Blood levels of disease markers
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 108 | 107
ng/mL
  Baseline | 0.0695 [0.020 to 0.513] | 0.0530 [0.020 to 0.568]
  Day 14 | 0.0410 [0.020 to 2.880] | 0.0340 [0.020 to 0.120]
  Day 28 | 0.0380 [0.020 to 0.246] | 0.0350 [0.020 to 1.840]

46. Secondary Outcome: Correlation of Time to Clinical Improvement With Quartiles of D-Dimer Blood Levels at Day 6
Description: Kaplan-Meier analyses were used to investigate a potential relationship between blood levels of D-Dimer and time to clinical improvement. Estimates of the clinical outcome were evaluated separately for patients within each of the four quartiles of D-Dimer levels at Day 6.
Time Frame: D-Dimer levels at Day 6; Clinical outcome: Day 0 to EoS (EoS = Day 27 up to Day 42)
Population: Safety analysis set consisting of all randomized patients who received at least one dose of IMP.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 100 | 101
days
  Q 1 (Min to 275 ng/mL D-Dimer): number analyzed (Participants) | 20 | 31
  Q 1 (Min to 275 ng/mL D-Dimer) | 13.8 [7.6 to 14.8] | 13.8 [13.7 to 13.8]
  Q 2 (275 to 450 ng/mL D-Dimer): number analyzed (Participants) | 33 | 17
  Q 2 (275 to 450 ng/mL D-Dimer) | 13.7 [12.0 to 13.9] | 13.8 [10.8 to 15.8]
  Q 3 (450 to 731 ng/mL D-Dimer): number analyzed (Participants) | 21 | 29
  Q 3 (450 to 731 ng/mL D-Dimer) | 13.8 [13.7 to 14.8] | 13.8 [13.0 to 14.8]
  Q 4 (731 ng/mL to Max D-Dimer): number analyzed (Participants) | 26 | 24
  Q 4 (731 ng/mL to Max D-Dimer) | 13.7 [12.0 to 14.0] | 13.8 [13.7 to 14.0]

47. Secondary Outcome: Changing in Log 10 Copies in Spontaneous Sputum and Nasopharyngeal Swab Samples at Various Time Points
Description: Virologic markers: Severe Acute Respiratory Syndrome Coronavirus Virus (SARS-CoV-2) Mean Viral Load - log10 Copies in Spontaneous Sputum and Nasopharyngeal Swab Samples: changing of SARS-CoV-2 Viral Load in patients on Days 6,14,28
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: Change in log10 copies
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 67 | 72
Change in log10 copies
  Day 2 | -10020591.1 (38272166.5) | -62534293.5 (380490492.5)
  Day 6 | -12849771.3 (49984377.5) | -84355538.5 (416667915.1)
  Day 14 | -13617000.9 (51579374.1) | -89534493.9 (429884542.5)
  Day 28 | -15195922.3 (54087022.5) | -44774028.6 (249373454.1)

48. Secondary Outcome: Mean Viral Load - log10 Copies in Spontaneous Sputum and Nasopharyngeal Swab Samples
Description: Virologic markers :Severe Acute Respiratory Syndrome Coronavirus Virus (SARS-CoV-2) mean viral load - log10 copies in spontaneous sputum and nasopharyngeal swab samples:
  Time course of SARS-CoV-2 viral load
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (Standard Deviation); unit: log10 Copies
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 78 | 77
log10 Copies
  Baseline | 10966569.9 (46215130.5) | 75572844.7 (389541813.1)
  Day 6 | 33277.7 (168585.9) | 581813.6 (3313425.6)
  Day 14 | 37642.6 (281630.2) | 483522.2 (3851254.5)
  Day 28 | 181.6 (673.9) | 369.7 (2133.1)

49. Secondary Outcome: Number of Participants With 2 Consecutive Negative SARS-CoV-2 Reverse Transcriptase Polymerase Chain Reaction Tests at Least 24 Hours Apart
Description: Virologic markers: Qualitative Virologic Clearance in Spontaneous Sputum and Nasopharyngeal Swab Samples (= 2 Consecutive Negative SARS-CoV-2 Reverse Transcriptase Polymerase Chain Reaction Tests at Least 24 Hours Apart)
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
Participants | 69 | 77

50. Secondary Outcome: Rate of Conversion to a Negative SARS-CoV-2 (Qualitative) Test
Description: Virologic markers: conversion to a negative SARS-CoV-2 (qualitative) test on Day 28.
Time Frame: on Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 100 | 98
Participants | 57 | 60

51. Secondary Outcome: Time to Conversion to a Negative SARS-CoV-2 (Qualitative) Test
Description: Virologic markers : Time to Conversion to a Negative SARS-CoV-2 (Qualitative) Test Throughout the study. Only patients with viral load measured from nasopharyngeal swab and results provided by the central laboratory (Covance) were included.Conversion to a negative SARS-CoV-2 status is only assumed if a negative test is confirmed by all available subsequent assessments. This means for Day 28/early termination visit no confirmation is needed.
  If no conversion to a negative status is documented, patients will be censored for survival analysis at the time of the last documented positive test result.
Time Frame: Throughout the Study (Day 0 to Day 28)
Measure: Mean (90% Confidence Interval); unit: days
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 100 | 98
days | 13.8 [12.8 to 14.1] | 14.0 [13.7 to 27.8]

52. Secondary Outcome: Interleukin (IL)-17
Description: The profiles of immune system biomarkers
Time Frame: Day 0, 6, 14 and Day 28
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 106 | 107
pg/mL
  Baseline | 5.860 (0.000) | 5.860 (0.000)
  Day 6 | 5.860 (0.000) | 5.885 (0.177)
  Day 14 | 5.924 (0.621) | 5.860 (0.000)
  Day 28 | 5.866 (0.058) | 5.892 (0.308)

53. Secondary Outcome: Interleukin (IL)-1ß
Description: The profiles of immune system biomarkers
Time Frame: Day 0, 6, 14 and Day 28
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 106 | 107
ng/L
  Baseline | 0.668 (0.159) | 0.654 (0.032)
  Day 6 | 1.014 (1.865) | 1.100 (2.165)
  Day 14 | 0.976 (1.955) | 0.862 (0.970)
  Day 28 | 0.984 (2.240) | 0.662 (0.076)

54. Secondary Outcome: Interleukin (IL)-6
Description: The profiles of immune system biomarkers
Time Frame: Day 0, 6, 14 and 28
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 106 | 107
ng/L
  Baseline | 6.217 (8.037) | 5.093 (6.438)
  Day 6 | 5.441 (14.271) | 8.435 (30.854)
  Day 14 | 7.697 (25.514) | 5.536 (26.081)
  Day 28 | 3.437 (14.317) | 1.468 (1.879)

55. Secondary Outcome: Interferon Gamma (IFNγ)
Description: The profiles of immune system biomarkers
Time Frame: Day 0, 6, 14 and 28
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 106 | 107
pg/mL
  Baseline | 94.364 (166.465) | 92.190 (153.798)
  Day 6 | 28.654 (90.127) | 24.141 (77.850)
  Day 14 | 10.469 (13.224) | 38.192 (150.623)
  Day 28 | 17.013 (33.762) | 14.452 (21.067)

56. Secondary Outcome: Tumor Necrosis Factor Alpha
Description: The profiles of immune system biomarkers
Time Frame: Day 0, 6, 14 and 28
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 106 | 107
ng/L
  Baseline | 3.084 (3.314) | 3.310 (5.071)
  Day 6 | 6.617 (21.461) | 8.020 (18.418)
  Day 14 | 7.974 (18.526) | 12.064 (12.064)
  Day 28 | 4.778 (9.293) | 3.717 (5.690)

57. Secondary Outcome: Immunoglobulin (Ig)A and/or IgG Antibodies Against SARS-CoV-2
Description: Proportion of patients with IgA and/or IgG antibodies against SARS-CoV-2on at different time point
Time Frame: Day 6, 14 and 28
Population: Not all 220 patients were negative for SARS-CoV-2 in nasopharyngeal samples analyzed by the central laboratory throughout the study. Patients, where the reported result for IgA and IgG antibodies is "limit", are considered as "negative" for analysis.
Measure: Number; unit: percent of patients
Arm/Group | IMU-838 | Placebo
Number analyzed (Participants) | 110 | 110
percent of patients
  Day 6: number analyzed (Participants) | 100 | 102
  Day 6 | 86.0 | 83.8
  Day 14: number analyzed (Participants) | 96 | 97
  Day 14 | 96.9 | 94.3
  Day 28: number analyzed (Participants) | 90 | 97
  Day 28 | 98.3 | 96.9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until Day 60 after randomization
Arm/Group | IMU-838 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/110 | 2/110
Serious Adverse Events (participants affected / at risk) | 2/110 | 4/110
Other Adverse Events (participants affected / at risk) | 79/110 | 65/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMU-838 (N=110) | Placebo (N=110)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — COVID-19 pneumonia
Thrombosis (Vascular disorders) | 0 | 1 — Deep vein thrombosis
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (Investigations) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMU-838 (N=110) | Placebo (N=110)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Bradycardia (Cardiac disorders) | 4 (6) | 7 (10)
Sinus bradycardia (Cardiac disorders) | 6 (6) | 5 (5)
Tachycardia (Cardiac disorders) | 7 (7) | 2 (2)
Hepatocellular injury (Hepatobiliary disorders) | 3 (4) | 7 (7)
Alanine aminotransferase increased (Investigations) | 5 (5) | 6 (6)
Glycosylated haemoglobin increased (Investigations) | 10 (10) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7) | 8 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 23 (24) | 13 (13)
Headache (Nervous system disorders) | 8 (9) | 5 (6)
Haematuria (Renal and urinary disorders) | 7 (7) | 4 (4)
Hypertension (Vascular disorders) | 6 (8) | 4 (8)
Hypertensive crisis (Vascular disorders) | 6 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT04379271/Prot_SAP_000.pdf